CLINICAL TRIAL: NCT04867954
Title: Development of 4D Flow MRI for Risk Stratification of Variceal Bleeding in Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0220; 1R01DK125783 (NIH); A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 9/9/25 (Other: HS-IRB UW Madison)
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis, Liver; Gastroesophageal Varices; Fontan Procedure
MeSH Terms: conditions — Liver Cirrhosis | interventions — Ensure Plus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- Healthy volunteers: 7 healthy participants will be recruited.
  Interventions: Other: Pre-clinical validation contrast enhanced MRI
- Patients with small, low-risk GEV: Patients with small, low-risk Gastroesophageal varices (GEV) will be recruited.
  Interventions: Other: Pre-clinical validation contrast enhanced MRI
- Patients with large, high-risk GEV: Patients with large, high-risk Gastroesophageal varices (GEV) will be recruited.
  Interventions: Other: Pre-clinical validation contrast enhanced MRI
- Patients scheduled for screening or surveillance esophagogastroduodenoscopy (EGD): 100 patients diagnosed with cirrhosis and scheduled for screening or surveillance esophagogastroduodenoscopy (EGD) procedure will be recruited. Participants will complete a single research visit, lasting approximately 2 hours, that will include the following procedures:
  * Participants will fast for 12 hours prior to arriving.
  * An IV will be placed and a blood sample collected (~11 mL, if necessary).
  * All participants will undergo research MRI lasting approximately 1.5 hours
  Interventions: Other: Ensure Plus®; Other: Clinical validation MRI
- Obese patients: 20 obese patients will be recruited
  Interventions: Other: Pre-clinical validation contrast enhanced MRI + fasting
- Participants with Fontan repair and diagnosed Fontal associated liver disease (FALD): 5 participants with Fontan repair and diagnosed FALD will be recruited.
  Interventions: Other: Ensure Plus®; Other: Clinical validation MRI

INTERVENTIONS:
Other: Ensure Plus® — In-between two MRI exams, patients will ingest a standardized meal of two cans (16oz) of Ensure Plus® (Abbott Laboratories), providing a 700cal meal (13g protein, 11g fat, 50g carbohydrates), proven to elicit a strong hyperemic splanchnic response.
  Groups: Participants with Fontan repair and diagnosed Fontal associated liver disease (FALD); Patients scheduled for screening or surveillance esophagogastroduodenoscopy (EGD)
Other: Pre-clinical validation contrast enhanced MRI — Participants will be asked to complete a single research visit that will include a contrast enhanced MRI scan lasting up to 1 hour. Participants will be asked to fast for at least 5 hours prior to the exam. Participants will be screened a final time for contraindications to contrast enhanced MR imaging; an IV will be placed; and participants will be positioned in the MR scanner, asked to lie as still as possible and to follow some breath hold instructions.
  Other Names: MRI
  Groups: Healthy volunteers; Patients with large, high-risk GEV; Patients with small, low-risk GEV
Other: Clinical validation MRI — Participants will be screened for any previous reactions to Ferumoxytol or GBCAs and dosing will be consistent with standard of care.
  Participants will then undergo a research MRI lasting approximately 1.5 hours.
  * All participants will be positioned in the MRI scanner for the initial scanning session (30 min) during which a 1/2 or 3/4 of the full dose of gadolinium based contrast agent (GBCA) or the total dose of Ferumoxytol will be administered.
  * The first 50 participants will be removed from the scanner bore, repositioned, and scanned for an additional 15 minutes (repeatability testing).
  * All participants will then be removed from the scanner and asked to consume 16 ounces of Ensure Plus®. After 20 minutes, they will be repositioned in the scanner for an additional scanning session (15 minutes) during which, the remaining 1/4 or 1/2 dose of GBCA will be administered, if required.
  Other Names: MRI
  Groups: Participants with Fontan repair and diagnosed Fontal associated liver disease (FALD); Patients scheduled for screening or surveillance esophagogastroduodenoscopy (EGD)
Other: Pre-clinical validation contrast enhanced MRI + fasting — Participants will be asked to complete a single research visit that will include a contrast enhanced MRI scan lasting up to 1.5 hours. Participants will be asked to fast for at least 5 hours prior to the exam. Participants will be screened a final time for contraindications to contrast enhanced MR imaging; an IV will be placed; and participants will be positioned in the MR scanner, asked to lie as still as possible and to follow some breath hold instructions.
  Other Names: MRI
  Groups: Obese patients

SUMMARY:
The goal of this research is to validate novel non-invasive Magnetic resonance imaging (MRI) biomarkers to detect Gastroesophageal varices (GEV) in patients with cirrhosis, including fractional flow change in the portal vein and elevated azygos flow.

End-stage liver disease (cirrhosis) is characterized by advanced fibrosis, liver failure, and portal hypertension. There are many causes of cirrhosis, including viral hepatitis, alcohol abuse, and perhaps most importantly, non-alcoholic fatty liver disease (NAFLD) and its aggressive subset, non-alcoholic steatohepatitis (NASH). 3 million new cases of end-stage liver disease (cirrhosis) are expected over the next decade. In cirrhosis, portosystemic collaterals that shunt blood away from the liver develop due to increased portal pressure. Gastroesophageal varices (GEV) are the most clinically relevant because they can cause fatal internal bleeding. GEV bleeding carries ~20% mortality at 6 weeks, and ~34% overall mortality. Identification of at-risk varices, prior to bleeding, is of paramount importance to initiate primary prophylaxis. To identify and treat at-risk patients, current guidelines recommend regular esophagogastroduodenoscopy (EGD) and variceal band ligation. Detection of high-risk GEV is key to initiating primary prophylaxis, which can reduce mortality by 50-70%.

However, endoscopy is invasive and often unnecessary when no treatment is required. Therefore, the American Association for the Study of Liver Diseases has identified the development of "non-invasive markers that predict the presence of high-risk varices" as a major unmet need.

DETAILED DESCRIPTION:
The overall goal of this research is to implement advanced non-invasive 4D flow MRI biomarkers to predict the presence of treatable but potentially lethal GEV in patients with cirrhosis. This would facilitate the triage of patients with high-risk GEV to therapeutic EGD, while reducing unnecessary EGD procedures in patients without them.

The primary biological mechanism for development of GEV is elevated portal pressure and reversal of flow in the left gastric vein (LGV). Applying 4D flow MRI, investigators aim to detect and quantify reversed flow in the LGV to detect GEV at risk for bleeding.

Aim 1: Perform pre-clinical validations of an optimized, accelerated radial 4D flow MRI strategy, and of fat mitigation strategies for radial 4D flow MRI.

Aim 2: Determine the diagnostic performance of radial 4D flow MRI, in cirrhotic adults including

1. diagnostic accuracy to identify high-risk GEV using EGD as reference standard, and
2. test-retest repeatability Aim 3: Evaluate the effects and added value of a meal challenge to assess for high-risk GEV.

Aim 4: Compare the accuracy of 4D flow MRI to current non-invasive markers of liver disease.

Aim 5: Determine the feasibility of radial 4D flow MRI in participants with FALD to detect differences in mesenteric response to a meal challenge when compared to healthy controls and participants with other types of liver disease.

Research Procedures

Pre-Clinical Validation (Phase 1): A total of 21 participants (7 healthy volunteers, 14 patients with GEV) to evaluate the optimized 4D flow methods, and 20 obese subjects to evaluate fat-mitigation strategies, will be enrolled. Participants will be asked to complete a single research visit that will include a contrast enhanced MRI scan lasting up to 1 hour. Participants will be asked to fast for at least 5 hours prior to the exam. Participants will be screening a final time for contraindications to contrast enhanced MR imaging; an IV will be placed; and participants will be positioned in the MR scanner, asked to lie as still as possible and to follow some breath hold instructions.

Clinical Validation (Phase 2-3): A total of 105 patients diagnosed with cirrhosis will be enrolled. Participants will be asked to complete a single research visit, lasting approximately 2 hours, that will include the following procedures:

* Participants will be asked to fast for 12 hours prior to arriving.
* An IV will be placed for tracer administration
* Participants will undergo a research MRI lasting approximately 1.5 hours (up to 1 hour of total scan time)

  * All participants will be positioned in the MRI scanner for the initial scanning session (30 min) during which the first dose of GBCA (3/4 of total dose) or the total dose of Ferumoxytol will be administered.
  * 50 participants will be removed from the scanner bore, repositioned, and scanned for an additional 15 minutes (repeatability testing).
  * All participants will then be removed from the scanner and asked to consume 16 ounces of Ensure Plus®. After 20 minutes, they will be repositioned in the scanner for an additional scanning session (15 min) during which, a second dose of GBCA (1/4 of total dose) will be administered if required.

ELIGIBILITY:
Inclusion Criteria for Aim 1:

* Healthy volunteers: Adults (>18 years) with no known liver pathology
* Obese volunteers: Adults (>18 years), no known liver pathology, body mass index (BMI) ≥ 35
* Patients: Adults (>18 years) with known cirrhosis and known Gastroesophageal varices

Exclusion Criteria for Aim 1:

* contraindications to MRI
* hypersensitivity reactions to both contrast agents
* patients with recent treatment for varices with embolization, TIPS, or other endovascular treatment
* patients with active GEV bleeding; known occlusive thrombus in portal vein, splenic vein, or superior mesenteric vein.
* patients with large HCC with known PC involvement.

Inclusion criteria for Aim 2-4:

* Adults (>18 years) with known cirrhosis scheduled for EGD to assess for GEV.

Exclusion Criteria for Aim 2-4:

* Contraindications to MRI
* Recent treatment (< 1 year) for varices
* Known occlusive thrombus in portal vein; splenic vein, or superior mesenteric vein
* Large hepatocellular carcinoma (HCC) with known PV involvement
* Hypersensitivity reactions to both contrast agents
* Participants requiring conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI scan will be allowed to participate as long as the following criteria are met:

  * The participant has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of the medication.
  * The participant comes to the research visit with a driver.

Inclusion Criteria for Aim 5:

* Adults (>18 years) with Fontan repair and diagnosed FALD

Exclusion Criteria for Aim 5:

* Contraindications to MRI
* Recent treatment (< 1 year) for varices
* Known occlusive thrombus in portal vein; splenic vein, or superior mesenteric vein
* Large hepatocellular carcinoma (HCC) with known PV involvement
* Hypersensitivity reactions to both contrast agents
* Participants requiring conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI scan will be allowed to participate as long as the following criteria are met:

  * The participant has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of the medication.
  * The participant comes to the research visit with a driver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For pre-clinical validation (Aim 1), a total of 21 participants will be recruited: 7 healthy volunteers, 14 patients with GEV. For clinical validation (Aim 2-4), 100 patients will be recruited from the UWHC endoscopy clinics. For Aim 5, 5 participants will be recruited from from the UWHC endoscopy clinics.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Receiver operation characteristic (ROC) curve analysis to determine diagnostic accuracy | 2 hours
  Receiver operation characteristic (ROC) curve analysis will be performed to determine the diagnostic accuracy of 4D flow MRI to differentiate high-risk GEV from absent or low-risk GEV. The area under the curve (AUC) will be estimated for each flow measurement with 95% confidence intervals. The primary analysis is based on fractional flow change in the portal vein.
Variation in postprandial flow after Meal Challenge | pre and post meal (approximately 2 hours)
  Variations in flow after a meal will be analyzed under(log-)linear mixed effects (LME) models.
Repeatability of 4D flow MRI: measured by summary measures of test-retest agreement with 95% Confidence intervals(CIs). | 2 hours
  Repeatability of all flow measurements and fractional flow changes will be measured using intra-class correlation coefficient (ICC), and the wishing-subject coefficient of variation (wCV) will be estimated as summary measures of test-retest agreement with 95% CIs.
Diagnostic accuracy of 4D Flow MRI to detect high-risk gastroesophageal varices (GEV) compared to esophagogastroduodenoscopy (EGD) as the reference standard | Baseline
  Sensitivity and specificity of fractional flow change in the portal vein (FFCPV) and azygos flow thresholds

SECONDARY OUTCOMES:
Aspartate aminotransferase-to-platelet ratio index (APRI) | Within 3 months
  APRI is a way for doctors to measure how healthy a patient's liver is when they have a liver disease.
  APRI = [(AST/upper limit of normal)/platelet count]x100
Fibrosis 4 (FIB-4) index | Within 3 months
  The Fibrosis-4 score helps to estimate the amount of scarring in the liver. FIB-4 = age (years) × AST [IU/L] / [platelet count × sqr(ALT [IU/L])]
Liver and spleen stiffness measurement by 2D spin-echo MR elastography | Within 3 months
  2D spin-echo MR elastography will be acquired to assess liver and spleen stiffness, using a single or dual-paddle system to ensure adequate wave-propagation in the liver and spleen
Liver proton density fat fraction (PDFF) as assessed by chemical shift encoded MRI (CSE-MRI) | Within 3 months
  Liver proton density fat fraction (PDFF) is a biomarker of hepatic steatosis. It will be measured by Chemical shift encoded MRI (CSE-MRI; IDEAL IQ, GE Healthcare),pioneered at UW-Madison. It will help characterizing the possible confounders affecting 4D flow MRI
Hepatic iron level quantitation by in vivo R2* MRI method | Within 3 months
  R2* is an imaging method used in MRI. R2* = (1/T2*) where R2* is a relaxation rate measured in units of Hz ([1/sec]). R2* is commonly used to look at iron levels by measuring the relaxation times of hydrogen nuclei affected by iron. The presence of the iron results in the shortening of proton relaxation times (T2*), thus increasing R2*. R2* will be measured by Chemical shift encoded MRI (CSE-MRI; IDEAL IQ, GE Healthcare), pioneered at University of Wisconsin (UW)-Madison. It will help characterizing the possible confounders affecting 4D flow MRI
Child-Turcotte-Pugh (CTP) score for prognosis of cirrhosis | Within 3 months
  The Child-Turcotte-Pugh (CTP) score is used to assess the severity of cirrhosis. Parameters included are Encephalopathy, Ascites, Bilirubin levels, Albumin levels, Prothrombin Time and International Normalized Ratio (PT/INR) . Parameters are scored on point 1-3. CTP score is obtained by adding the score for each parameter. CTP scores can be categorized into A= 5-6 points, B=7-9 points and C=10-15 points. Higher points correspond to more severe cirrhosis state.
Repeatability of 4D Flow MRI measurements in cirrhotic patients | Two hours
  Intraclass correlation coefficient (ICC) for flow measurements
Feasibility of radial 4D Flow MRI and meal challenge protocol in FALD patients | Two hours
  Completion rate and image quality scores
Postprandial mesenteric and portal flow response in FALD vs cirrhosis and healthy controls | pre and post meal (approximately 2 hours)
  Absolute and fractional flow changes in portal and mesenteric vessels

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reeder, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No